CLINICAL TRIAL: NCT02641353
Title: A Phase 1, Open-Label, Randomized Three-Period, Six-Sequence Crossover Study In Healthy Adult Subjects To Evaluate The Bioavailablity Of An Oral Suspension Formulation Relative To The Tablet Formulation Of Apremilast And To Assess The Effect Of Food On The Pharmacokinetics Of The Oral Suspension Formulation
Brief Title: Study to Evaluate Bioavailability of Apremilast Oral Suspension Relative to Tablet and to Assess Effect of Food on the Pharmacokinetics (PK) of the Oral Suspension
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CC-10004-CP-032; 20200157 (Other: Amgen Study ID)
Expanded Access: NCT03740516 (No longer available)
Record Dates: First submitted 2015-12-23; First posted 2015-12-29 (Estimated); Results first posted 2021-08-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: Healthy Volunteers
Keywords: Apremilast; Healthy volunteers; Bioavailability; Food effect; Pharmacokinetic
MeSH Terms: interventions — apremilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A: Apremilast 30 mg Tablet - Fasted (Experimental): A single oral dose of 30 mg apremilast tablet after an overnight fast.
  Interventions: Drug: Apremilast Tablet
- Treatment B: Apremilast 30 mg Oral Suspension - Fasted (Experimental): A single oral dose of 30 mg apremilast oral suspension formulation (6 mL) after an overnight fast.
  Interventions: Drug: Apremilast Oral Suspension
- Treatment C - Apremilast 30 mg Oral Suspension - Fed (Experimental): A single oral dose of 30 mg apremilast oral suspension formulation (6 mL) after a high-fat meal.
  Interventions: Drug: Apremilast Oral Suspension

INTERVENTIONS:
Drug: Apremilast Tablet — 30 mg tablet
  Other Names: Otzela; CC-10004
  Arms: Treatment A: Apremilast 30 mg Tablet - Fasted
Drug: Apremilast Oral Suspension — 30 mg oral suspension
  Other Names: Otzela; CC-10004
  Arms: Treatment B: Apremilast 30 mg Oral Suspension - Fasted; Treatment C - Apremilast 30 mg Oral Suspension - Fed

SUMMARY:
The purpose of this study is to assess how much of apremilast is found in the blood unchanged when administered as an oral suspension compared to when it is administered as a tablet formulation. The effect of food on apremilast oral suspension will also be evaluated. In addition, information on the safety and tolerability of apremilast will be obtained.

DETAILED DESCRIPTION:
This is a phase 1, open-label, randomized, three-period, six-sequence crossover study in healthy subjects. The study will consist of a screening phase, baseline (Day -1), three study periods, and a follow-up phone call. Each study period will be four days in duration (Day 1 through Day 4) followed by a five-day washout between doses.

Eligible participants will be admitted into the study center on Day -1 of study Period 1 for baseline measurements. During each study period, participants will receive a single 30 mg oral dose of apremilast on Day 1 according to the assigned treatment sequence. Participants will be confined at the study center from Day 1 of study Period 1 through Day 4 of study Period 3, including the 5 day washout between doses. All participants will be discharged from the study center on Day 4 of study Period 3 following completion of required study procedures. A follow-up phone call will occur approximately four days after the discharge from the study center.

The study will be conducted in compliance with International Conference on Harmonisation (ICH) Good Clinical Practices (GCPs).

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy ALL of the following criteria to be eligible for enrollment into the study:

1. Must understand and voluntarily sign a written Informed Consent (ICF) prior to any study-related procedures being performed.
2. Must be able to communicate with the investigator, understand and comply with the requirements of the study, and agree to adhere to restrictions and examination schedules.
3. Male and female subjects of any race between 18 to 55 years of age (inclusive), and in good health as determined by the Investigator at the time of signing the informed consent document.
4. Have a Body Mass Index (BMI) between 18 and 33 kg/m^2 (inclusive).
5. No clinically significant laboratory test results as determined by the investigator.
6. At the screening visit, must be afebrile, with supine systolic blood pressure (BP): 90 to 140 mmHg, supine diastolic BP: 50 to 90 mmHg, and pulse rate: 40 to 110 bpm. Eligibility criteria for vital signs performed during check-in and/or predose on Day 1 will be at the discretion of the Investigator.
7. Must have a normal or clinically acceptable 12-lead electrocardiogram (ECG). Subjects must have a QTcF value ≤ 450 msec.
8. Contraception Requirements:

   * Must comply with the following acceptable forms of contraception. All female of childbearing potential (FCBP) must use one of the approved contraceptive options as described below while taking apremilast and for at least 28 days after administration of the last dose of the apremilast.
   * At the time of study entry, and at any time during the study when a FCBP's contraceptive measures or ability to become pregnant changes, the Investigator will educate the subject regarding contraception options and the correct and consistent use of effective contraceptive methods in order to successfully prevent pregnancy

   All FCBP must have a negative pregnancy test at Visits 1 and 2. All FCBP subjects who engage in activity in which conception is possible must use one of the approved contraceptive options described below:

   Option 1: Any one of the following highly effective methods: hormonal contraception (oral, injection, implant, transdermal patch, vaginal ring); intrauterine device (IUD); tubal ligation; or partner's vasectomy; OR Option 2: Male or female condom (latex condom or non-latex condom NOT made out of natural [animal] membrane [for example, polyurethane]); PLUS one of the following additional barrier methods: (a) diaphragm with spermicide; (b) cervical cap with spermicide; or (c) contraceptive sponge with spermicide.

   Male subjects (including those who have had a vasectomy) who engage in activity in which conception is possible must use barrier contraception (latex or non-latex condoms NOT made out of natural [animal] membrane [for example, polyurethane]) while on investigational product (IP) and for at least 28 days after the last dose of IP.
9. Must agree to refrain from donating sperm, blood or plasma (other than for this study) while participating in this study and for at least 28 days after the last dose of investigational product.
10. Subject is willing and able to adhere to the study visit schedule and other protocol requirements

Exclusion Criteria:

The presence of ANY of the following will exclude any healthy subject from enrollment into the study:

1. History of any clinically significant and relevant neurological, psychiatric, gastrointestinal, renal, hepatic, cardiovascular, psychological, pulmonary, metabolic, endocrine, hematological, allergic disease, drug allergies, or other major disorders.
2. Any condition which places the subject at unacceptable risk if he were to participate in the study, or confounds the ability to interpret data from the study.
3. Use of any prescribed systemic or topical medication within 30 days of the first dose administration.
4. Use of any non-prescribed systemic or topical medication (including vitamin/mineral supplements, and herbal medicines) within 14 days of the first dose administration, Any surgical or medical condition possibly affecting drug absorption, distribution, metabolism and excretion, eg, bariatric procedure, colon resection, irritable bowel syndrome, Crohn's disease, etc. Subjects with cholecystectomy and appendectomy may be included.
5. Exposure to an investigational drug (new chemical entity) within 30 days prior to the first dose administration or 5 half-lives of that investigational drug, if known (whichever is longer).
6. Donated blood or plasma within 8 weeks before the first dose administration to a blood bank or blood donation center.
7. History of drug abuse (as defined by the current version of the Diagnostic and Statistical Manual [DSM]) within 2 years before dosing, or a positive drug screen reflecting consumption of illicit drugs.
8. History of alcohol abuse (as defined by the current version of the DSM) within 2 years before dosing, or a positive alcohol screen.
9. Known to have hepatitis, or known to be a carrier of the hepatitis B surface antigen (HBsAg), or hepatitis C antibody (HCV Ab), or have a positive result to the test for HBsAg, HCV Ab, or human immunodeficiency virus (HIV) antibodies at Screening.

   -

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2016-01-05 (Actual); Primary Completion 2016-02-27 (Actual); Study Completion 2016-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- Covance Clinical Research Unit Inc, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at a single site in the United States. The study consisted of three treatment periods separated by a 5-day washout period.
Pre-assignment Details: Participants were randomly assigned to one of six treatment sequences. On day 1 of each treatment sequence participants received one of the following according to their assigned treatment sequence:
  * Treatment A: Single oral dose of 30 mg apremilast tablet under fasted conditions
  * Treatment B: Single oral dose of 30 mg apremilast oral suspension formulation under fasted conditions
  * Treatment C: Single oral dose of 30 mg apremilast oral suspension formulation under fed conditions
Groups:
- Sequence 1: Treatments ACB: Participants received 30 mg apremilast oral tablet after an overnight fast on day 1 of treatment period 1, 30 mg apremilast oral suspension after a high-fat meal on day 1 of treatment period 2, and 30 mg apremilast oral suspension after an overnight fast on day 1 of treatment period 3.
- Sequence 2: Treatments CBA: Participants received 30 mg apremilast oral suspension after a high-fat meal on day 1 of treatment period 1, 30 mg apremilast oral suspension after an overnight fast on day 1 of treatment period 2, and 30 mg apremilast oral tablet after an overnight fast on day 1 of treatment period 3.
- Sequence 3: Treatments BAC: Participants received 30 mg apremilast oral suspension after an overnight fast on day 1 of treatment period 1, 30 mg apremilast oral tablet after an overnight fast on day 1 of treatment period 2, and 30 mg apremilast oral suspension after a high-fat meal on day 1 of treatment period 3.
- Sequence 4: Treatments ABC: Participants received 30 mg apremilast oral tablet after an overnight fast on day 1 of treatment period 1, 30 mg apremilast oral suspension after an overnight fast on day 1 of treatment period 2, and 30 mg apremilast oral suspension after a high-fat meal on day 1 of treatment period 3.
- Sequence 5: Treatments CAB: Participants received 30 mg apremilast oral suspension after a high-fat meal on day 1 of treatment period 1, 30 mg apremilast oral tablet after an overnight fast on day 1 of treatment period 2, and 30 mg apremilast oral suspension after an overnight fast on day 1 of treatment period 3.
- Sequence 6: Treatments BCA: Participants received 30 mg apremilast oral suspension after an overnight fast on day 1 of treatment period 1, 30 mg apremilast oral suspension after a high-fat meal on day 1 of treatment period 2, and 30 mg apremilast oral tablet after an overnight fast on day 1 of treatment period 3.
Period: Overall Study
Arm/Group | Sequence 1: Treatments ACB | Sequence 2: Treatments CBA | Sequence 3: Treatments BAC | Sequence 4: Treatments ABC | Sequence 5: Treatments CAB | Sequence 6: Treatments BCA
Started | 5 | 5 | 6 | 6 | 6 | 6
Completed | 5 | 5 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Participants received a single dose of the following three treatments in one of six treatment sequences:
  * Treatment A: Single oral dose of 30 mg apremilast tablet under fasted conditions
  * Treatment B: Single oral dose of 30 mg apremilast oral suspension formulation under fasted conditions
  * Treatment C: Single oral dose of 30 mg apremilast oral suspension formulation under fed conditions
Arm/Group | Total
Number analyzed (Participants) | 34
Age, Continuous [Mean (Full Range); unit: years] | 33.3 [19 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Black or African American | 14
  White | 17
  Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Apremilast
Description: Concentrations of apremilast in plasma were measured using a validated liquid chromatography tandem mass spectrometry assay.
Time Frame: Predose and at 0.5, 1, 1.5, 2, 3, 5, 8, 12, 24, 36, 48, 60 and 72 hours after dosing on day 1 of each treatment period.
Population: The pharmacokinetic (PK) population included all participants who received at least one dose of apremilast and had at least one measurable concentration datum.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Treatment C: Apremilast 30 mg Oral Suspension - Fed: A single oral dose of 30 mg apremilast oral suspension formulation (6 mL) after a high-fat meal.
Arm/Group | Treatment A: Apremilast 30 mg Tablet - Fasted | Treatment B: Apremilast 30 mg Oral Suspension - Fasted | Treatment C: Apremilast 30 mg Oral Suspension - Fed
Number analyzed (Participants) | 34 | 34 | 34
ng/mL | 323 (34.5) | 274 (32.2) | 215 (33.7)
Statistical Analysis 1: Comparison: Treatment A: Apremilast 30 mg Tablet - Fasted vs Treatment B: Apremilast 30 mg Oral Suspension - Fasted; To assess the bioavailability between the apremilast oral suspension and tablet formulation an analysis of variance (ANOVA) model, with treatment, sequence, and period as fixed effects and subject nested within sequence as a random effect, was performed on the natural log-transformed Cmax; Test type: Other; Geometric Mean Ratio = 84.9, 90% CI 2-sided [77.3 to 93.2] — Ratio of adjusted geometric means (Treatment B / Treatment A) expressed as a percentage
Statistical Analysis 2: Comparison: Treatment B: Apremilast 30 mg Oral Suspension - Fasted vs Treatment C: Apremilast 30 mg Oral Suspension - Fed; To assess the effect of food on the PK of apremilast oral suspension formulation, an ANOVA model, with treatment, sequence, and period as fixed effects and subject nested within sequence as a random effect, was performed on the natural log-transformed Cmax; Test type: Other; Geometric Mean Ratio = 78.2, 90% CI 2-sided [71.2 to 86.0] — Ratio of adjusted geometric means (Treatment C / Treatment B) expressed as a percentage

2. Primary Outcome: Area Under the Concentration-time Curve From Time Zero to the Last Measured Time Point (AUC0-t) for Apremilast
Description: Concentrations of apremilast in plasma were measured using a validated liquid chromatography tandem mass spectrometry assay. AUC from time zero to the last measured time point was calculated by the linear trapezoidal method.
Time Frame: Predose and at 0.5, 1, 1.5, 2, 3, 5, 8, 12, 24, 36, 48, 60 and 72 hours after dosing on day 1 of each treatment period.
Population: The pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Treatment A: Apremilast 30 mg Tablet - Fasted | Treatment B: Apremilast 30 mg Oral Suspension - Fasted | Treatment C: Apremilast 30 mg Oral Suspension - Fed
Number analyzed (Participants) | 34 | 34 | 34
ng*h/mL | 3130 (38.9) | 2740 (43.1) | 3160 (41.3)
Statistical Analysis 1: Comparison: Treatment A: Apremilast 30 mg Tablet - Fasted vs Treatment B: Apremilast 30 mg Oral Suspension - Fasted; To assess the bioavailability between the apremilast oral suspension and tablet formulation an ANOVA model, with treatment, sequence, and period as fixed effects and subject nested within sequence as a random effect, was performed on the natural log-transformed AUC0-t; Test type: Other; Geometric Mean Ratio = 87.6, 90% CI 2-sided [83.0 to 92.5] — Ratio of adjusted geometric means (Treatment B / Treatment A) expressed as a percentage
Statistical Analysis 2: Comparison: Treatment B: Apremilast 30 mg Oral Suspension - Fasted vs Treatment C: Apremilast 30 mg Oral Suspension - Fed; To assess the effect of food on the PK of apremilast oral suspension formulation, an ANOVA model, with treatment, sequence, and period as fixed effects and subject nested within sequence as a random effect, was performed on the natural log-transformed AUC0-t; Test type: Other; Geometric Mean Ratio = 115.3, 90% CI 2-sided [109.2 to 121.7] — Ratio of adjusted geometric means (Treatment C / Treatment B) expressed as a percentage

3. Primary Outcome: Area Under the Concentration-time Curve From Time Zero to Infinity (AUC0-∞) for Apremilast
Description: Concentrations of apremilast in plasma were measured using a validated liquid chromatography tandem mass spectrometry assay. AUC from time zero to infinity was calculated as (AUC0-t + Ct/λz), where Ct is the last quantifiable concentration, and λz is the apparent terminal rate constant.
Time Frame: Predose and at 0.5, 1, 1.5, 2, 3, 5, 8, 12, 24, 36, 48, 60 and 72 hours after dosing on day 1 of each treatment period.
Population: The pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Treatment A: Apremilast 30 mg Tablet - Fasted | Treatment B: Apremilast 30 mg Oral Suspension - Fasted | Treatment C: Apremilast 30 mg Oral Suspension - Fed
Number analyzed (Participants) | 34 | 34 | 34
ng*h/mL | 3160 (38.7) | 2760 (43.2) | 3190 (41.3)
Statistical Analysis 1: Comparison: Treatment A: Apremilast 30 mg Tablet - Fasted vs Treatment B: Apremilast 30 mg Oral Suspension - Fasted; To assess the bioavailability between the apremilast oral suspension and tablet formulation an ANOVA model, with treatment, sequence, and period as fixed effects and subject nested within sequence as a random effect, was performed on the natural log-transformed AUC0-∞; Test type: Other; Geometric Mean Ratio = 87.8, 90% CI 2-sided [83.2 to 92.6] — Ratio of adjusted geometric means (Treatment B / Treatment A) expressed as a percentage
Statistical Analysis 2: Comparison: Treatment B: Apremilast 30 mg Oral Suspension - Fasted vs Treatment C: Apremilast 30 mg Oral Suspension - Fed; To assess the effect of food on the PK of apremilast oral suspension formulation, an ANOVA model, with treatment, sequence, and period as fixed effects and subject nested within sequence as a random effect, was performed on the natural log-transformed AUC0-∞; Test type: Other; Geometric Mean Ratio = 115.0, 90% CI 2-sided [109.0 to 121.7] — Ratio of adjusted geometric means (Treatment C / Treatment B) expressed as a percentage

4. Primary Outcome: Time to Maximum Observed Plasma Concentration (Tmax) of Apremilast
Description: as for outcome 1
Time Frame: Predose and at 0.5, 1, 1.5, 2, 3, 5, 8, 12, 24, 36, 48, 60 and 72 hours after dosing on day 1 of each treatment period.
Population: The PK population
Measure: Median (Full Range); unit: hours
Arm/Group | Treatment A: Apremilast 30 mg Tablet - Fasted | Treatment B: Apremilast 30 mg Oral Suspension - Fasted | Treatment C: Apremilast 30 mg Oral Suspension - Fed
Number analyzed (Participants) | 34 | 34 | 34
hours | 2.00 [1.00 to 5.00] | 2.00 [1.50 to 5.00] | 5.00 [1.50 to 12.00]
Statistical Analysis 1: Comparison: Treatment A: Apremilast 30 mg Tablet - Fasted vs Treatment B: Apremilast 30 mg Oral Suspension - Fasted; Tmax was analyzed by nonparametric methods. The median difference and 90% confidence interval (CI) of the median difference were calculated from the Hodges-Lehrmann estimate; Test type: Other; p = 0.1508, Wilcoxon signed-rank test; Median Difference = 0.25, 90% CI 2-sided [0.00 to 0.50] — Median difference (Treatment B - Treatment A) calculated from the Hodges-Lehmann estimate
Statistical Analysis 2: Comparison: Treatment B: Apremilast 30 mg Oral Suspension - Fasted vs Treatment C: Apremilast 30 mg Oral Suspension - Fed; Tmax was analyzed by nonparametric methods. The median difference and 90% CI of the median difference were calculated from the Hodges-Lehrmann estimate; Test type: Other; p < 0.0001, Wilcoxon signed-rank test; Median Difference = 2.25, 90% CI 2-sided [1.27 to 3.25] — Median difference (Treatment C - Treatment B) calculated from the Hodges-Lehmann estimate

5. Primary Outcome: Terminal Elimination Half-life (T1/2) of Apremilast
Time Frame: Predose and at 0.5, 1, 1.5, 2, 3, 5, 8, 12, 24, 36, 48, 60 and 72 hours after dosing on day 1 of each treatment period.
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Treatment A: Apremilast 30 mg Tablet - Fasted | Treatment B: Apremilast 30 mg Oral Suspension - Fasted | Treatment C: Apremilast 30 mg Oral Suspension - Fed
Number analyzed (Participants) | 34 | 34 | 34
hours | 7.89 (34.5) | 8.51 (31.8) | 7.54 (30.8)

6. Primary Outcome: Apparent Clearance of Apremilast From Plasma After Extravascular Administration (CL/F)
Time Frame: Predose and at 0.5, 1, 1.5, 2, 3, 5, 8, 12, 24, 36, 48, 60 and 72 hours after dosing on day 1 of each treatment period.
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Treatment A: Apremilast 30 mg Tablet - Fasted | Treatment B: Apremilast 30 mg Oral Suspension - Fasted | Treatment C: Apremilast 30 mg Oral Suspension - Fed
Number analyzed (Participants) | 34 | 34 | 34
L/h | 9.51 (38.7) | 10.9 (43.2) | 9.42 (41.3)

7. Primary Outcome: Apparent Volume of Distribution of Apremilast During the Terminal Phase (Vz/F)
Time Frame: Predose and at 0.5, 1, 1.5, 2, 3, 5, 8, 12, 24, 36, 48, 60 and 72 hours after dosing on day 1 of each treatment period.
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Treatment A: Apremilast 30 mg Tablet - Fasted | Treatment B: Apremilast 30 mg Oral Suspension - Fasted | Treatment C: Apremilast 30 mg Oral Suspension - Fed
Number analyzed (Participants) | 34 | 34 | 34
L | 108 (45.2) | 133 (43.7) | 102 (38.9)

8. Primary Outcome: Lag Time (Tlag) of Apremilast
Description: Lag time is the delay between the time of administration and start of absorption.
Time Frame: Predose and at 0.5, 1, 1.5, 2, 3, 5, 8, 12, 24, 36, 48, 60 and 72 hours after dosing on day 1 of each treatment period.
Population: PK population
Measure: Median (Full Range); unit: hours
Arm/Group | Treatment A: Apremilast 30 mg Tablet - Fasted | Treatment B: Apremilast 30 mg Oral Suspension - Fasted | Treatment C: Apremilast 30 mg Oral Suspension - Fed
Number analyzed (Participants) | 34 | 34 | 34
hours | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]

9. Primary Outcome: Relative Bioavailability (F) of Apremilast Oral Suspension Formulation
Description: Relative bioavailability of the oral suspension formulation compared to the tablet formulation, calculated as (AUC0-∞/Dose[oral suspension]) / (AUC0-∞/Dose[tablet]) * 100%.
Time Frame: Predose and at 0.5, 1, 1.5, 2, 3, 5, 8, 12, 24, 36, 48, 60 and 72 hours after dosing on day 1 of each treatment period.
Population: PK population. Relative bioavailability calculated for each of the oral suspension treatments as pre-specified in the Protocol.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percent availability
Arm/Group | Treatment B: Apremilast 30 mg Oral Suspension - Fasted | Treatment C: Apremilast 30 mg Oral Suspension - Fed
Number analyzed (Participants) | 34 | 34
percent availability | 87.6 (16.1) | 101 (14.3)

10. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events
Description: An adverse event (AE) is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a participant during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the participant's health, including laboratory test values, regardless of etiology.
  A treatment-emergent AE (TEAE) was defined as any AE that occurred after dosing of the study drug.
  A serious adverse event (SAE) is any AE occurring at any dose that:
  * Resulted in death;
  * Was life-threatening;
  * Required inpatient hospitalization or prolongation of existing hospitalization;
  * Resulted in persistent or significant disability/incapacity;
  * Was a congenital anomaly/birth defect;
  * Constituted an important medical event.
Time Frame: From first dose of study drug in treatment period 1 to 8 days after the last dose; up to 18 days.
Population: The safety population included all participants who received at least one dose of apremilast.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: Apremilast 30 mg Tablet - Fasted | Treatment B: Apremilast 30 mg Oral Suspension - Fasted | Treatment C: Apremilast 30 mg Oral Suspension - Fed
Number analyzed (Participants) | 34 | 34 | 34
Participants
  Any treatment-emergent adverse event (TEAE) | 8 | 10 | 6
  TEAEs related to study drug | 4 | 7 | 4
  Serious adverse events | 0 | 0 | 0
  TEAEs leading to discontinuation | 0 | 0 | 0
  TEAEs leading to death | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug in treatment period 1 to 8 days after the last dose; up to 18 days.
Arm/Group | Treatment A: Apremilast 30 mg Tablet - Fasted | Treatment B: Apremilast 30 mg Oral Suspension - Fasted | Treatment C: Apremilast 30 mg Oral Suspension - Fed | Total
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/34 | 0/34 | 0/34
Other Adverse Events (participants affected / at risk) | 5/34 | 10/34 | 3/34 | 15/34
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A: Apremilast 30 mg Tablet - Fasted (N=34) | Treatment B: Apremilast 30 mg Oral Suspension - Fasted (N=34) | Treatment C: Apremilast 30 mg Oral Suspension - Fed (N=34) | Total (N=34)
Constipation (Gastrointestinal disorders) | 0 | 2 | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 5 | 1 | 5
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Flatulence (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Nausea (Gastrointestinal disorders) | 2 | 2 | 0 | 4
Feeling hot (General disorders) | 0 | 2 | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2
Headache (Nervous system disorders) | 2 | 2 | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.